CLINICAL TRIAL: NCT04551417
Title: DoVe Trial: a Randomized Controlled Trial Comparing Dorsal Onlay Versus Ventral Onlay in Isolated Bulbar Urethral Strictures
Brief Title: DoVe Trial: Dorsal Onlay Versus Ventral Onlay in Isolated Bulbar Urethral Strictures
Acronym: DoVe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC-06890
Record Dates: First submitted 2020-06-29; First posted 2020-09-16 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Urethra Stenosis
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dorsal onlay graft urethroplasty (Active Comparator)
  Interventions: Procedure: Free graft urethroplasty
- Ventral onlay graft urethroplasty (Experimental)
  Interventions: Procedure: Free graft urethroplasty

INTERVENTIONS:
Procedure: Free graft urethroplasty — Free graft urethroplasty will be performed either with ventral or dorsal onlay of the graft.

SUMMARY:
For bulbar urethral strictures, it remains unclear whether ventral onlay graft urethroplasty is non-inferior to dorsal onlay graft urethroplasty in terms of patency rates.

DETAILED DESCRIPTION:
Urethral stricture disease is a common urological condition in men. Although rigorous epidemiologic data is sparse, the existing papers report an incidence varying between 0.6 and 1.4 percent1. Urethral strictures can occur throughout the entire length of the urethra, but mainly involve the anterior urethra and, in particular, the bulbar segment2.

The International Consultation on Urologic Diseases (ICUD) recommends anastomotic repair (AR) urethroplasty for isolated, short, bulbar urethral strictures3. However, AR urethroplasty is only possible up to a certain point of stricture length. The elasticity of the bulbar urethra is estimated to be about 25% and given the average bulbar urethral length of 10 cm, one could simply calculate that strictures up to 2.5 cm can be treated with AR urethroplasty. However, this border of 2.5 cm is rather arbitrary as additional length may be gained through the different maneuvers of Webster et al., enabling the option of AR for even longer strictures4. Furthermore, the location of the stricture within the bulbar segment plays an important role as well: a proximal bulbar stricture location allows AR for longer strictured segments (> 2.5 cm) than a more distal stricture location which nears the penoscrotal angle. Anyhow, the key for a successful AR procedure is to perform a well-vascularized and tension-free anastomosis5. Whenever this is impossible to achieve, even after performing the length-gaining maneuvers of Webster et al., it is recommended to perform a so-called 'substitution urethroplasty' in which the strictured area of the urethra is opened and augmented with a free graft or a pedicled flap5.

Within the option of substitution urethroplasty, free graft urethroplasty (FGU) definitely represents the easiest and most straightforward treatment option. Herein, urethral surgeons initially started by placing grafts ventrally 'on' the urethra: 'ventral onlay FGU'. Later, Barbagli et al. started placing grafts dorsally: 'dorsal onlay FGU'6. They advocated that this dorsal graft position would lead to better graft anchorage, less graft mobility and less graft sacculation. However, to date, there is no indisputable data to support the choice of one technique over another, not from a surgical point of view, nor from a functional point of view7. Furthermore, studies investigating this issue are mostly retrospective and thus only entail a low level of evidence7.

Against this background, the aim of the DoVe trial is to directly compare dorsal onlay and ventral onlay FGU for both surgical and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations (Appendix B).
* Age ≥ 18 years.
* Male patient.
* Fit for operation, based on the surgeon's expert opinion.
* Isolated bulbar urethral stricture confirmed by imaging.
* Preputium, penile shaft skin, buccal mucosa and lingual mucosa are allowed as free graft material in the executed dorsal onlay or ventral onlay FGU.
* Patient is able and willing to attend the follow-up consultations.

Exclusion Criteria:

* Absence of signed written informed consent (Appendix B).
* Age < 18 years.
* Female patients.
* Transgender patients.
* Patients unfit for operation.
* Concomitant urethral strictures at other urethral locations (penile urethra, membranous urethra, prostatic urethra, bladder neck).
* A unique urethral stricture at other urethral locations (penile urethra, membranous urethra, prostatic urethra, bladder neck).
* Prior bulbar urethroplasty.
* Lichen Sclerosus related strictures.
* Strictures after failed hypospadias repair.
* Patients with neurogenic bladder.
* History of pelvic radiation therapy.
* Shift of technique to any other technique than dorsal or ventral onlay FGU due to any circumstance (post-hoc exclusion).
* Utilization of free graft material other than preputium, penile shaft skin, buccal mucosa or lingual mucosa.
* Any condition or situation, which, in the investigator's opinion, puts the patient at significant risk, could confound the study results, or may interfere significantly with the patient's participation in the study.
* Patient declares that it will be impossible for him to attend the follow-up consultations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival after 24 months | 24 months
  Failure is defined as the inability to pass a flexible 16 Fr cystoscope through the reconstructed area without damaging the urethral mucosa.

SECONDARY OUTCOMES:
Change in postoperative erectile function | Baseline questionnaire, followed by questionnaire at 3, 12 and 24 months of follow-up.
  Assessed with IIEF 5 questionnaire (international index on erectile function: score between 5 and 25, higher scores indicating better erectile function)
Change in ejaculatory function | Baseline questionnaire, followed by questionnaire at 3, 12 and 24 months of follow-up.
  Assessed with MSHQ-EjD short form questionnaire (male sexual health questionnaire - ejaculatory dysfunction short form: score between 1 and 15, higher scores indicating better ejaculatory function)
Change in LUTS | Baseline question, followed by question at 3, 12 and 24 months of follow-up.
  Assessed with Peeling's voiding picture (score between 1 and 4, lower scores indicating better strength of the urinary stream)
Change in LUTS | Baseline questionnaire, followed by questionnaire at 3, 12 and 24 months of follow-up.
  Assessed with ICIQ-MLUTS module (international consultation on incontinence questionnaire - male lower urinary tract symptoms: score between 0 and 24, higher scores indicating more LUTS)
Change in urinary continence | Baseline questionnaire, followed by questionnaire at 3, 12 and 24 months of follow-up.
  Assessed with ICIQ-UI short form questionnaire (international consultation on incontinence questionnaire - urinary incontinence: score between 0 and 21, higher scores indicating more urinary incontinence)
Change in maximum flow rate | Uroflowmetry at baseline, followed by uroflowmetry at 3, 12 and 24 months of follow-up.
  Assessed with uroflowmetry (Qmax)
Change in quality of life | Baseline questionnaire, followed by questionnaire at 3, 12 and 24 months of follow-up.
  Assessed with EQ-5D-3L (5 questions on quality of life resulting in digit score, e.g. 11231, higher scores indicating worse quality of life)
Change in quality of life | Baseline questionnaire, followed by questionnaire at 3, 12 and 24 months of follow-up.
  Assessed with EQ-VAS (EQ-visual analogue scale: scale between 0 and 100, higher scores indicating better quality of life)
Patient satisfaction | Assessed after 3, 12 and 24 months of follow-up.
  Assessed with two general patient satisfaction questions
Postoperative complication rate | Within 90 days postoperatively
  Categorized according to the Clavien-Dindo classification system

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, Principal Investigator — University Hospital, Ghent; Wesley Verla, Study Director — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No